CLINICAL TRIAL: NCT02302612
Title: Multi-Component Behavioral Intervention for Complex Patients With CVD Risk. The Changing Results: Engage and Activate to Enhance Wellness (CREATE Wellness) Study
Brief Title: The CREATE Wellness Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CN-13-1672-H; R01HL117939 (NIH)
Record Dates: First submitted 2014-11-21; First posted 2014-11-27 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Diabetes; Heart Disease; Hypertension; Dyslipidemia
Keywords: chronic conditions; complex patients; engagement; activation
MeSH Terms: conditions — Diabetes Mellitus; Heart Diseases; Hypertension; Dyslipidemias; Chronic Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CREATE Wellness (Experimental): Patients allocated to the intervention arm will receive three group sessions with between visit contacts designed to increase activation and engagement with their care plans. They will also continue to be enrolled in the KP PHASE disease management program.
  Interventions: Behavioral: CREATE Wellness
- Usual Care Control (Active Comparator): Patients allocated to the control arm will continue to receive usual care, including disease management within the KP PHASE program.
  Interventions: Other: Usual Care Control

INTERVENTIONS:
Behavioral: CREATE Wellness — Patients allocated to the intervention arm will receive three group sessions with between visit contacts designed to increase activation and engagement with their care plans. They will also continue to be enrolled in the KP PHASE program
  Arms: CREATE Wellness
Other: Usual Care Control — Patients allocated to the control arm will continue to receive usual care, including disease management within the KP PHASE program.
  Arms: Usual Care Control

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of death in the U.S. Efforts to improve CVD risk factors often fall short in complex patients with multiple co-morbid conditions, a growing, expensive, and high-risk segment of the U.S. population. The investigators are testing a multi-component behavioral intervention designed to help complex patients with CVD and other concurrent chronic conditions to become more effective agents of their own care.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of death in the U.S. Despite the availability of evidence-based guidelines and efficacious therapies, however, many patients do not achieve the full benefit of CVD risk reduction. In particular, complex patients (defined as those patients who do not respond to current disease management approaches) with multiple concurrent chronic conditions represent a key segment of the population that would benefit from new approaches to care. In response to PA-12-024: Behavioral Interventions to Address Multiple Chronic Conditions in Primary Care, which seeks "practical interventions…to modify behaviors using a common approach" among patients with multiple co-morbidities, the investigators are testing an integrated behavioral intervention designed to improve a core set of chronic disease self-management skills and to overcome common barriers to care engagement encountered by this increasingly important segment of the U.S. adult primary care population. This randomized trial will be conducted within Kaiser Permanente Northern California (KPNC), an integrated care delivery system serving over 3.2 million members, including patients insured through Medicare and state Medicaid programs. The investigators will evaluate the intervention in 3 KPNC primary care practices by enrolling 576 complex patients who have persistently (≥ 2 years) uncontrolled CVD risk factors (e.g. hypertension, hyperlipidemia, diabetes) despite being enrolled in a CVD disease management program. This behavioral intervention is designed to activate and engage patients, identify potentially hidden barriers to care such as alcohol misuse or sub-clinical depression, and to develop individualized care plans that are designed to catalyze more effective primary care management. Randomization will be at the patient-level. The investigators will examine the impact of the intervention on clinical outcomes (control of systolic blood pressure, HbA1c (if with diabetes), statin treatment rates) after 12 months and patient-reported outcomes (patient activation, medication adherence, and mental health status) after 6 months. By focusing on core health skills and care barriers, this patient-focused intervention seeks to enable complex patients to become more effective agents of their own care and to thereby achieve similar clinical benefits as less complex patients.

ELIGIBILITY:
Inclusion Criteria:

* Kaiser Permanente Northern California members enrolled in the PHASE disease management program and not meeting all goals of care for the preceding 2 years.

Exclusion Criteria:

* Schizophrenia or personality disorder
* Unable to communicate in English
* Unwilling to participate in group-based in-person program
* Pregnant
* Terminal or debilitating illness

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 647 (Actual)
Dates: Start 2015-01; Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Composite CVD Goal | 12-months
  We will compare the proportion of patients in the two study arms who achieve all three clinical goals of the PHASE disease management program (blood pressure control, HbA1c control (if applicable), and statin prescription) 12 months after enrollment. Risk factor control is defined according to the PHASE disease management program protocol.

SECONDARY OUTCOMES:
Perceived efficacy in patient-physician interactions (PEPPI) - 10 items | 6 months
  We will compare proportion of patients with improvement between baseline and follow-up PEPPI 10-item survey scores between study arms
Effective Consumer Scale (EC-17) | 6 months
  We will compare proportion of patients with improvement between baseline and follow-up EC-17 scores between study arms
Patient Activation Measure (PAM) - 13 items | 6 months
  We will compare proportion of patients with improvement between baseline and follow-up PAM scores between study arms

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Grant, MD MPH, Principal Investigator — Division of Research, KPNC
Locations (1):
- Kaiser Permanente San Jose Sabrina Wood, BA (510) 891-3551 Sabrina.B.Wood@kp.org, San Jose, California, United States

REFERENCES:
- [Derived] Iturralde E, Sterling SA, Uratsu CS, Mishra P, Ross TB, Grant RW. Changing Results-Engage and Activate to Enhance Wellness: A Randomized Clinical Trial to Improve Cardiovascular Risk Management. J Am Heart Assoc. 2019 Dec 3;8(23):e014021. doi: 10.1161/JAHA.119.014021. Epub 2019 Nov 30. PMID 31787053
- [Derived] Torres DX, Lu WY, Uratsu CS, Sterling SA, Grant RW. Knowing How to Ask Good Questions: Comparing Latinos and Non-Latino Whites Enrolled in a Cardiovascular Disease Prevention Study. Perm J. 2019;23:18-258. doi: 10.7812/TPP/18-258. PMID 30939290
- [Derived] Miller-Rosales C, Sterling SA, Wood SB, Ross T, Makki M, Zamudio C, Kane IM, Richardson MC, Samayoa C, Charvat-Aguilar N, Lu WY, Vo M, Whelan K, Uratsu CS, Grant RW. CREATE Wellness: A multi-component behavioral intervention for patients not responding to traditional Cardiovascular disease management. Contemp Clin Trials Commun. 2017 Oct 4;8:140-146. doi: 10.1016/j.conctc.2017.10.001. eCollection 2017 Dec. PMID 29696203